CLINICAL TRIAL: NCT05116085
Title: A Single-Arm, Multicenter, Open-Label, Phase 2 Study to Investigate the Efficacy and Safety of Tislelizumab (BGB-A317) as Neo-Adjuvant Treatment in Patients With Early-Stage (Stage II-III) Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) Colorectal Cancer
Brief Title: Efficacy and Safety of Tislelizumab (BGB-A317) as Neo-Adjuvant Treatment in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-214; CTR20212779 (Other: ChinaDrugTrials)
Record Dates: First submitted 2021-10-20; First posted 2021-11-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab (Experimental): Tislelizumab administered intravenously before surgery during the neo-adjuvant phase
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Administered intravenously
  Other Names: BGB-A317

SUMMARY:
This study will evaluate the safety, and tolerability of neo-adjuvant treatment with tislelizumab in participants with early-stage (Stage II-III) Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG Performance status of 0 or 1.
2. Pathologically (histologically) confirmed diagnosis of potentially resectable Stage II or Stage III Colon/Rectal Cancer (CRC) with MSI-H confirmed by sponsor designated central laboratory or known MSI-H status by local laboratory. Participants should be eligible for an R0 resection with curative intent.
3. Evaluable or measurable disease as assessed by the investigator per RECIST v1.1.
4. Adequate hematologic and organ function, defined by protocol-specified laboratory test results, obtained within 7 days before first dose.

Exclusion Criteria:

1. Any prior therapy for current CRC, including chemotherapy or radiotherapy or immunotherapy.
2. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days before first dose.
3. Active autoimmune diseases or history of autoimmune diseases that may relapse.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Major pathological response (MPR) rate | approximately 16 months
  MPR rate is defined as the percentage of participants with ≤ 10% residual viable tumor in the resected primary tumor

SECONDARY OUTCOMES:
Pathological complete response (pCR) rate | approximately 16 months
  Percentage of participants with absence of residual tumor
Event-free survival (EFS) | approximately 50 months
  Time from first dose until disease progression
2-year/3-year EFS rate | approximately 50 months
  Percentage of participants free from EFS events at 2 years and 3 years estimated using the Kaplan-Meier method.
Proportion of participants expressing Potential Biomarkers in Blood | approximately 50 months
  Potential biomarkers include immune cell infiltration, PD-L1 expression, tumor mutational burden (TMB) and DNA mutation, gene expression profile (GEP)
Number of Participants With Clinically Significant Laboratory Values | approximately 16 months
  Laboratory parameters include hematology , chemistry, coagulation and urinalysis
Number of Participants With Clinically Significant Vital Signs | approximately 16 months
  Vital signs include pulse rate and blood pressure
Number of Participants With Clinically Significant Physical Examination Findings | approximately 16 months
  A full physical examination includes head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal and musculoskeletal systems
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | approximately 16 months
  Number of participants with one or more TEAE, including serious adverse events and immune-mediated adverse events, graded according to NCI-CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University Branch South, Qingdao, Shandong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/